CLINICAL TRIAL: NCT00548392
Title: Sonographic Visibility of Breast Biopsy Marker Clips Up to 4 Weeks After Placement
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Ethicon Endo-Surgery (Industry); GE Healthcare (Industry)
Responsible Party: Peter Eby, University of Washington/SCCA
Other Study IDs: 6263
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer
Keywords: breast; cancer; ultrasound; high risk; marker clip
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — none/not applicable
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine how long collagen based marker clips remain visible by ultrasound after placement in suspicious breast lesions and if collagen based marker clips can be reliably identified in the operating room and serve as effective guidance for surgical removal of high risk or malignant breast lesions.

DETAILED DESCRIPTION:
Many breast cancers and other breast lesions are discovered as a palpable abnormality by patients or their providers during a breast exam. Diagnostic imaging and biopsy of these lesions may reveal high-risk or malignant findings. These palpable lesions can be removed in the operating room by the surgeon using touch as guidance. However, there are many lesions discovered by screening examinations that surgeons cannot palpate. When this occurs, a radiologist will percutaneously place a wire or wires at the site of the breast lesion using sonographic or mammographic guidance. The surgeon then uses the wires as a guide for complete and successful resection of the lesion.

New marker devices have been developed that are sonographically visible. They consist of the standard mammographically visible metallic clip surrounded by a sonographically visible collagen plug. It is hypothesized that radiologists and surgeons can effectively localize the clip with intra-operative ultrasound and then resect the lesion. If so, the pre-operative wire localization procedure could be eliminated. This could improve the patient experience while saving time and money by reducing the number of invasive procedures from 3 (biopsy, wire-localization and operation) to 2 (biopsy and operation).

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicious breast lesions that have undergone biopsy and marker clip placement within 28 days (4 weeks) of pre-operative consultation visit.
* Patients or their legal representative must be able to provide written informed consent.
* Patients must be over 18 years old.

Exclusion Criteria:

* Under the age of 18 years
* Unable to give written informed consent
* Patients will be excluded if the clip was placed more than 4 weeks prior to their pre-operative appointment or wire-localization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Visibility of marker clip after placement in suspicious breast lesions. | Within 4 weeks of placement

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Eby, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States